CLINICAL TRIAL: NCT00148174
Title: Predictors and Intervention for Noncompliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9611M11943; 2P01DK013083-40A1 (NIH)
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Kidney Transplantation
Keywords: Medication adherence; Patient compliance; Kidney transplant; Organ rejection; Allograft loss; Drug monitoring
MeSH Terms: conditions — Medication Adherence; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phone calling (Experimental): Phone calling to encourage improved adherence
  Interventions: Behavioral: Intensive telephone followup

INTERVENTIONS:
Behavioral: Intensive telephone followup — Telephone calling

SUMMARY:
This is a randomized controlled intervention trial in poorly compliant patients, testing whether improved compliance behavior decreases rates of acute rejection risk and graft loss.

Hypothesis: A study of an intensive intervention focused on the least compliant patients and beginning 3 months post-transplant. Effective intervention will reduce the number of acute rejection episodes and thus the occurrence of chronic rejection and graft loss.

DETAILED DESCRIPTION:
Our original studies demonstrated "early" noncompliant behavior predicted adverse transplantation outcomes including acute graft rejection and graft loss. In this study, we are randomly assigning a telephone intervention in a prospective cohort of medically noncompliant patients. Standard therapy includes specifically warning patients about the risks of noncompliant behavior, and the formal intervention is randomized so half of these patients will also receive intensive telephone followup, intended to improve medication compliance and reduce adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant
* Discharged from hospital with functioning graft

Exclusion Criteria:

* Risk of recurrent primary renal disease, e.g. hemolytic uremic syndrome, oxalosis, membranoproliferative glomerulonephritis type II, focal,segmental glomerulosclerosis with nephrotic syndrome
* Patients with active psychosis
* Patients not using azathioprine, sirolimus, or mycophenolate mofetil for immunosuppression at the time of discharge
* Patients taking the liquid form of azathioprine or mycophenolate mofetil
* Patients who are younger than 14 yrs. old
* Patients who do not speak English
* Receiving extra-renal organ except for pancreas,either simultaneously or previously
* Patients who live and will be followed outside of the United States, except Canada
* Patients who are physically unable to open the Medication Event Monitoring System(MEMS)cap
* Patients who are not responsible for taking their own medications, e.g. living in a medical care facility

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 1998-08; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Graft loss | prospective

SECONDARY OUTCOMES:
Acute rejection | prospective
Death | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Nevins, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States